CLINICAL TRIAL: NCT06239480
Title: SELVA: A Multicenter, Phase 3 Baseline-Controlled Study Evaluating the Safety and Efficacy of QTORIN 3.9% Rapamycin Anhydrous Gel in the Treatment of Microcystic Lymphatic Malformations
Brief Title: SELVA: A Phase 3 Study Evaluating QTORIN 3.9% Rapamycin Anhydrous Gel in the Treatment of Microcystic Lymphatic Malformations
Acronym: SELVA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALV-09
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Microcystic Lymphatic Malformation
Keywords: Lymphangioma circumscriptum; Lymphatic malformation; Vascular malformation; Topical; Sirolimus; Rapamycin; Congenital malformation; Non-infective disorder of lymphatic vessels and lymph nodes
MeSH Terms: conditions — Lymphangioma; Lymphatic Abnormalities; Vascular Malformations; Congenital Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental)
  Interventions: Drug: QTORIN 3.9% Rapamycin Anhydrous Gel

INTERVENTIONS:
Drug: QTORIN 3.9% Rapamycin Anhydrous Gel — QTORIN 3.9% Rapamycin Anhydrous Gel

SUMMARY:
SELVA: A Multicenter, Phase 3 Baseline-Controlled Study Evaluating the Safety and Efficacy of QTORIN 3.9% Rapamycin Anhydrous Gel in the Treatment of Microcystic Lymphatic Malformations

The main purpose of this study is to assess the change in microcystic lymphatic malformations IGA after 24 weeks of treatment with QTORIN 3.9% Rapamycin Anhydrous Gel in approximately 40 participants with microcystic lymphatic malformations. Efficacy will be evaluated at 24 weeks and patients have the option of continuing on treatment for >24 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must be at least 3 years of age at time of consent/assent
* Participant must have a clinically confirmed superficial/cutaneous microcystic lymphatic malformation

Key Exclusion Criteria:

* Participants who have vascular malformations that interfere with evaluating the target microcystic lymphatic malformation
* Participants with complicated vascular anomalies with severe systemic symptoms that require systemic therapy
* The participant's treatment area is mainly in any wet mucosa or within the orbital rim
* Participants who are pregnant or planning to become pregnant

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall microcystic lymphatic malformations Investigator Global Assessment (mLM-IGA) | At Week 24
  A multi-point scale with higher values indicating improvement.

SECONDARY OUTCOMES:
Change in the blinded clinician microcystic lymphatic malformations Multicomponent Severity Scale (mLM-MCSS) | At Week 24
  A multi-point scale with lower values indicating improvement.
Change in the live clinician microcystic lymphatic malformations Multicomponent Severity Scale (mLM-MCSS) | Change from Baseline to Week 24
  A multi-point scale with lower values indicating improvement.
Overall patient global impression of change (PGI-C) | Change from Baseline to Week 24
  A multi-point scale with lower values indicating improvement.
Change in Overall Clinician Global Impression of Severity (CGI-S) | Change from Baseline to Week 24
  A multi-point scale with lower values indicating improvement.
Change in Overall Patient Global Impression of Severity (PGI-S) | Change from Baseline to Week 24
  A multi-point scale with lower values indicating improvement.
Incidence and severity of adverse events | From Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Teng, Principal Investigator — Stanford University
Locations (15):
- United States (15):
  - Children's Hospital of Orange County, Irvine, California
  - Stanford University, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Vascular Birthmark Institute, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas, Dell Children's, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah